CLINICAL TRIAL: NCT02168608
Title: Remote Ischemia Precondition for Hepatic Protection in Patients Undergoing Hepatectomy: A Single-center Randomized Controlled Trial
Brief Title: Remote Ischemia Precondition (RIPC) for Hepatic Protection in Patients Undergoing Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Wei-feng Yu, professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EHBHKY2013-003-006
Record Dates: First submitted 2014-06-11; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Liver Neoplasms
Keywords: hepatic ischemia reperfusion injury; ischemia precondition; remote ischemia precondition; anti-inflammation
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemia precondition (Experimental): patients in this arm accepted RIPC procedure after induction of anesthesia
  Interventions: Other: Remote ischemia precondition
- None remote ischemia precondition (Experimental): patients in this arm didn't accept RIPC procedure after induction of anesthesia
  Interventions: Other: None remote ischemia precondition

INTERVENTIONS:
Other: Remote ischemia precondition — Three cycles of 5-min ischemia/5-min reperfusion induced by a blood pressure cuff placed on the right upper arm served as RIPC stimulus.
  Arms: Remote ischemia precondition
Other: None remote ischemia precondition — Placed an uninflated cuff on the right upper arm for 30 min.
  Arms: None remote ischemia precondition

SUMMARY:
Remote ischemia precondition could protect the liver from ischemia reperfusion injury in patients undergoing hepatectomy.

DETAILED DESCRIPTION:
Remote ischemia precondition (RIPC) had been proofed beneficial to ischemia reperfusion injury of heart, kidney, liver, brain and spinal cord in experimentation on animals. And the clinical studies of RIPC were mainly focused on heart, RIPC's protection effect on hepatic ischemia reperfusion injury in patients undergoing hepatectomy still remains unknown, So we designed this study to demonstrate the hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* No other main organ diseases, American society of Anesthesiologists (ASA) classification Ⅰ-Ⅱ grade
* Selective hepatectomy, one time hepatic portal occlusion
* Child-Pugh A

Exclusion Criteria:

* Peripheral vessels diseases
* Not the same surgical procedure as expected
* Administered anti-inflammatory drugs as glucocorticoid etc
* Diagnosed of diabetes
* History of liver surgery
* History of hepatic interventional therapy, radiofrequency therapy,radiotherapy and chemotherapy
* Refuse to join the research
* Patients with psychopathy
* Acute infection need antibiotic therapy
* Hepatic artery or portal vein embolism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
survival rate | 30 days postoperatively

SECONDARY OUTCOMES:
alanine aminotransferase (ALT) level in patients' blood | 1 day postoperatively
  Examine the patients's blood sample for ALT level at 1 day postoperatively
aspartic transaminase (AST) level in patients' blood | 1 day postoperatively
  Examine the patients's blood sample for AST level at 1 day postoperatively
alanine aminotransferase (ALT) level in patients' blood | 3 days postoperatively
  Examine the patients's blood sample for ALT level at 3 days postoperatively
aspartic transaminase (AST) level in patients' blood | 3 days postoperatively
  Examine the patients's blood sample for AST level at 3 days postoperatively
alanine aminotransferase (ALT) level in patients' blood | 7 days postoperatively
  Examine the patients's blood sample for ALT level at 7 days postoperatively
aspartic transaminase (AST) level in patients' blood | 7 days postoperatively
  Examine the patients's blood sample for AST level at 7 days postoperatively
complications | 30 days postoperatively
  Number of participants with adverse events within 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, professor, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Kin H, Zhao ZQ, Sun HY, Wang NP, Corvera JS, Halkos ME, Kerendi F, Guyton RA, Vinten-Johansen J. Postconditioning attenuates myocardial ischemia-reperfusion injury by inhibiting events in the early minutes of reperfusion. Cardiovasc Res. 2004 Apr 1;62(1):74-85. doi: 10.1016/j.cardiores.2004.01.006. PMID 15023554
- [Background] Huguet C, Addario-Chieco P, Gavelli A, Arrigo E, Harb J, Clement RR. Technique of hepatic vascular exclusion for extensive liver resection. Am J Surg. 1992 Jun;163(6):602-5. doi: 10.1016/0002-9610(92)90567-b. PMID 1595841
- [Background] Delva E, Camus Y, Nordlinger B, Hannoun L, Parc R, Deriaz H, Lienhart A, Huguet C. Vascular occlusions for liver resections. Operative management and tolerance to hepatic ischemia: 142 cases. Ann Surg. 1989 Feb;209(2):211-8. doi: 10.1097/00000658-198902000-00012. PMID 2916865
- [Background] Clavien PA, Yadav S, Sindram D, Bentley RC. Protective effects of ischemic preconditioning for liver resection performed under inflow occlusion in humans. Ann Surg. 2000 Aug;232(2):155-62. doi: 10.1097/00000658-200008000-00001. PMID 10903590
- [Background] Azoulay D, Lucidi V, Andreani P, Maggi U, Sebagh M, Ichai P, Lemoine A, Adam R, Castaing D. Ischemic preconditioning for major liver resection under vascular exclusion of the liver preserving the caval flow: a randomized prospective study. J Am Coll Surg. 2006 Feb;202(2):203-11. doi: 10.1016/j.jamcollsurg.2005.10.021. PMID 16427543